CLINICAL TRIAL: NCT02722213
Title: Mindfulness-Based Stress Reduction as an Adjunct Intervention to Cardiac Rehabilitation: A Pilot Study
Brief Title: Mindfulness & Stress Management Study for Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Fairview Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1603M85502
Record Dates: First submitted 2016-03-10; First posted 2016-03-29 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Heart Diseases; Heart Failure; Myocardial Infarction; Chronic Stable Angina; Coronary Artery Bypass; Angioplasty
MeSH Terms: conditions — Heart Diseases; Heart Failure; Myocardial Infarction; Angina, Stable | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): The intervention is an 8-week Mindfulness-Based Stress Reduction (MBSR) course, with 8 weekly 2.5-hour group sessions, and 1 all-day (6.5 hours) retreat, taught per standard protocol in a group setting. The course includes instruction and practice of meditation, breathing techniques, gentle yoga and Tai Chi poses, with shared discussion, brief readings and home practice between sessions. Participants will continue with usual care and receive standard educational materials on healthy lifestyles and stress management.
  Note: This study will recruit patients eligible for exercise-based cardiac rehabilitation (CR). Randomization to either MBSR or control (no MBSR) condition will occur within two strata (CR; no CR) will occur based on current enrollment in CR at time of study enrollment.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR).
- Control (No MBSR) (No Intervention): Those randomized to the control condition will continue with usual care and receive standard educational materials on healthy lifestyles and stress management. At the end of the study control participants will receive a compact disc and workbook on MBSR.
  Note: This study will recruit patients who are eligible for traditional exercise-based cardiac rehabilitation (CR). Randomization will be stratified based on whether or not patients are actively enrolled in CR at the time of the study. Within each stratum, participants will be randomized to either the intervention (MBSR) or control (no MBSR) condition.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR). — MBSR is a combination of mindfulness meditation, breathing practices, gentle yoga, and other relaxation techniques; it is taught in a manualized 8-week program, does not require special equipment, and can be practiced safely by people of all abilities
  Arms: Mindfulness-Based Stress Reduction

SUMMARY:
The guideline-recommended standard of care for patients who have experienced a heart attack, heart failure, or other coronary event or procedure is exercise-based cardiac rehabilitation (CR). Despite proven benefits, traditional CR is severely underutilized. Moreover, what is typically lacking from traditional CR programs is effective psychosocial risk management. This represents a critical gap in care given the well-documented psychosocial needs of this patient population.The objective of this feasibility study is to conduct a pilot randomized controlled trial (RCT) of Mindfulness-Based Stress Reduction (MBSR) versus usual care in CR-eligible cardiac patients. Randomization will be stratified within two strata based on participation in CR (yes/no) among CR-eligible patients. The primary goals of this pilot study are to: 1) obtain estimates of treatment effects and variability; 2) evaluate recruitment and retention strategies; and 3) examine the safety of the MBSR protocol in CR-eligible patients.

DETAILED DESCRIPTION:
Objectives:

The objective of this feasibility study is to conduct a pilot randomized controlled trial (RCT) of Mindfulness-Based Stress Reduction (MBSR) versus usual care in CR-eligible cardiac patients. Randomization will be stratified within two strata based on participation in CR (yes/no) among CR-eligible patients. The primary goals of this pilot study are to: 1) obtain estimates of treatment effects and variability; 2) evaluate recruitment and retention strategies; and 3) examine the safety of the MBSR protocol in CR-eligible patients.

Design and Outcomes:

The study design is a randomized controlled trial with randomization in two strata. The primary outcome will be a change (improvement) in heart rate variability (HRV) as assessed by a 24-hour Holter monitor worn by patients three times throughout the study: (pre- and post-intervention and 9-month follow-up). Time domain variables SDNN (the standard deviation of R-to-R intervals and RMSSD (the root mean square of successive differences in adjacent R-to-R intervals will be assessed. Time domain variables will be assessed via 24-hour Holter monitoring at baseline, 3-month follow-up and 9-month follow-up. HRV is a well-established method to assess the autonomic nervous system. Secondary outcomes will include psychosocial measures (depressive symptoms, mentally unhealthy days, stress, and anxiety) as well as cardiovascular risk factors (systolic blood pressure, body mass index, high density lipoprotein cholesterol, triglycerides, hemoglobin A1C, and c-reactive protein). All participants will undergo a baseline assessment, followed by randomization to the treatment or control condition, and three follow-up assessments, at 3, 6, and 9 months after randomization. The 3-month follow-up will occur immediately post-intervention and the 9-month follow up will occur 6-months post-intervention. The baseline, 3-month and 9-month (final) follow-up assessments will be in-person and will include questionnaires on stress and emotions, quality of life, a short physical performance battery, a blood draw to assess lipids, high sensitivity C-Reactive Protein and hemoglobin A1c as well as the 24-hour Holter monitor to assess HRV. The 6-month follow-up assessment will be by telephone only and include brief assessments of moods, stress, and symptoms. The investigators anticipate the pilot study will be completed in 18 months.

Interventions and Duration:

Upon enrollment, participants will be randomized into two groups, the intervention group (MBSR) or the control group (no MBSR). Randomization will occur separately for those enrolled in CR and those not enrolled in CR. For those in the stratum that attends CR, the control condition will consist of CR only and usual care, whereas for participants in the stratum that does not attend CR, the control condition will consist of usual care. All participants in both strata will received standard printed materials on healthy lifestyles and stress management. The intervention lasts for 8 weeks and will occur within the first 12 weeks (3 months) after randomization. The standard outpatient Phase II CR program offered within the Fairview Hospital system is a traditional exercise-based program that includes an intake visit and up to 24 1-hour monitored exercise sessions (1-3 times per week for 8-24 weeks, individualized to patient needs and therapy goals) and up to 8 or 9 1-hour educational sessions. Patients participating in CR who are randomized to the intervention group will participate in the same standard outpatient Phase II CR as those individuals randomized to the control condition within this stratum, plus an 8-week MBSR course. The MBSR course is taught per a standard protocol in a group setting and consists of eight 2.5-hour weekly sessions and one 6.5-hour retreat; the MBSR course will be led by trained facilitators from the University of Minnesota Center for Spirituality and Healing.

Sample Size and Population:

The targeted enrollment is 48 participants, with 32 randomized to participate in MBSR across the two strata and 16 randomized to the control condition (no MBSR) who will receive usual care (this includes CR for those who have opted to enroll in CR). The investigators will recruit CR-eligible cardiac patients from three sites within the Fairview Hospital system that offer CR (Ridges in Burnsville, Southdale in Edina, and University of Minnesota Riverside Campus in Minneapolis), as well as through electronic health records, clinic visits with health care providers, advertisement and flyers located at clinics and the CR locations, and inclusion of the study on www.studyfinder.umn.edu.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 21 and older that are medically eligible and been referred for traditional exercise-based CR (heart attack within the past 12 months, open heart surgery such as coronary bypass/valve/heart transplant, coronary angioplasty or stent placement, current stable angina, or heart failure)
* Willing to participate in all assessments and be randomized to either study condition
* Able to give informed consent.

Exclusion Criteria:

* Has a cardiac pacemaker and is pacemaker-dependent or has an untreated atrial arrhythmia;
* Previously completed an MBSR course;
* Unable to read and write in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change (improvement) in heart rate variability (HRV). | 0-9 months
  Time domain and frequency domain variables will be assessed via 24-hour Holter monitoring at baseline, 3-month follow-up and 9-month follow-up. HRV is a well-established method to assess the autonomic nervous system, and has been shown to be a predictor of hard outcomes in cardiac patients. Given the deranged autonomic milieu in these patients, HRV is an appropriate surrogate end point for improved outcomes in this cohort.

SECONDARY OUTCOMES:
Psychosocial function | 0-9 months
  Depressive symptoms, anxiety, stress, and health-related quality of life measures will be used to assess psychosocial function at baseline and changes in psychosocial function over the course of the study.
Cardiovascular risk factors: C-reactive protein (CRP), lipids, hemoglobin A1c (HgA1c) | 0-9 months
  Measures of lipids, inflammation (CRP) and glucose metabolism (HgA1c) will be obtained at 3 time points (baseline; 3-month follow-up; 9-month follow-up) to determine changes over the course of the study in these important cardiovascular risk factors.
Physical functioning | 0-9 months
  The Short Physical Performance Battery (SPPB) will be administered at baseline, 3-month follow-up and 9-month follow-up and will allow study investigators to evaluate changes in participants' physical function over time.

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Everson-Rose, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT02722213/Prot_SAP_000.pdf